CLINICAL TRIAL: NCT05011981
Title: Hemostatic Activity Following Left Atrial Appendage Occlusion
Brief Title: Hemostatic Activity Following LAAO
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Hemo-LAAO
Record Dates: First submitted 2021-08-12; First posted 2021-08-18 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Atrial Fibrillation; Stroke
MeSH Terms: conditions — Atrial Fibrillation; Stroke | interventions — Left Atrial Appendage Closure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Left Atrial Appendage Occlusion — Interventional left atrial appendage occlusion with the Amulet or Watchman device
  Other Names: Left Atrial Appendage Closure

SUMMARY:
The primary objective of this study is to prospectively investigate hemostatic activity following transcatheter left atrial appendage occlusion (LAAO).

DETAILED DESCRIPTION:
This is a prospective cohort study of patients undergoing transcatheter LAAO at Aarhus University Hospital. Hemostatic consequences following device implantation will be evaluated using blood samples collected pre- and post-procedurally, and serially during three months follow-up in 135 LAAO patients. Platelet function and characteristics, overall activation of the extrinsic coagulation pathway and the intrinsic contact activation pathway, as well as endothelial response to implantation, will be assessed through a wide range of biochemical analyses. Patients will serve as their own controls, with a final control blood sample collected at three-months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Atrial fibrillation (paroxysmal, persistent, or permanent)
* Admitted and eligible for LAAO
* Signed written consent

Exclusion Criteria:

* Known hereditary bleeding disorders (i.e. Hemophilia A and B, Von Willebrand disease)
* Platelet count < 75 x 109/ml

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Only patients already eligible for LAAO will be screened by clinical personnel and potentially recruited for participation. Blood samples will be systematically sampled during planned follow-up timepoints.
Sampling Method: Probability Sample
Enrollment: 135 (Estimated)
Dates: Start 2021-10-11 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change in coagulation activity | 7 days, 14 days, 90 days
  Coagulation activity as measured by prothrombin fragment 1+2

SECONDARY OUTCOMES:
Change in platelet activity | 7 days, 14 days, 90 days
  Incl. platelet count, turnover, and aggregation
Additional measures of changes in coagulation and contact activation | 7 days, 14 days, 90 days
  Incl. thrombin generation, fibrinogen, d-dimer and coagulation factors
Change in endothelial activation and response | 7 days, 14 days, 90 days
  Incl. changes in soluble thrombomodulin, syndecan-1, selectin and von Willebrand factor
Non-procedural bleeding events | 7 days, 14 days, 90 days
  As defined by the Bleeding Academic Research Consortium
Radiographical evidence of device endothelization | 7 days, 14 days, 90 days
  On CT indicated by no contrast patency distal to the LAAO device.
Radiographically confirmed device-related thrombosis | 7 days, 14 days, 90 days
  Defined as high grade HAT on follow-up cardiac CT or TEE

CONTACTS AND LOCATIONS:
Overall Officials: Anders Kramer, MD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus N, Central Denmark, Denmark